CLINICAL TRIAL: NCT05724056
Title: Comparison of the Efficacy and Safety of Idroflog® (Sodium Hyaluronate and Hydrocortisone) and Sodium Hyaluronate for the Treatment of Dry Eye Disease
Brief Title: Idroflog® for Treatment of Dry Eye Disease (IDROFLOG)
Acronym: IDROFLOG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alfa Intes Industria Terapeutica Splendore s.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-A01171-42
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye; Idroflog; Ocular
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled equally and randomly into either treatment group: Idroflog® or Sodium Hyaluronate 0.18% (Vismed®). Once randomized, participants will receive the intervention for 90 days, and will be followed up at 30 days, 60 days, and 90 days.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In order to maintain the blinding of the Investigator and his team, both products will be placed into identical boxes ("blinding-box"), identified only by a randomization number, without any indication of product identity or randomization arm.
  Each patient will be randomly assigned a randomization number, allocating him/her to either Idroflog® or Sodium Hyaluronate 0.18% (1:1) in accordance with a central randomisation table generated using a validated computer-program. Randomisation will be stratified per center and performed using a permuted random block design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Idroflog® (Experimental): Patients randomized in this group will be treated with Sodium Hyaluronate 2 mg/ml and Hydrocortisone 10 μg/ml.
  Interventions: Device: Idroflog®
- Sodium Hyaluronate 0.18% (Vismed®) (Active Comparator): Patients randomized in this group will be treated with Sodium Hyaluronate 0.18%.
  Interventions: Device: Sodium Hyaluronate 0.18% (Vismed®)

INTERVENTIONS:
Device: Idroflog® — The study intervention posology will be based on current labeling of Idroflog®. Participants will be self-administering one drop in each eye 4 times a day every day during the study period.
  Administration should follow the label guidelines. Participants should detach a single vial from the strip, remove the flap at the top by rotating it and instill 1 drop into the conjunctival sac of each eye, dropping them from above.
  Other Names: Study intervention
  Arms: Idroflog®
Device: Sodium Hyaluronate 0.18% (Vismed®) — The control intervention posology will be based on current labeling of Idroflog®. Participants will be self-administering one drop in each eye 4 times a day every day during the study period.
  Administration should follow the label guidelines. Participants should detach a single vial from the strip, remove the flap at the top by rotating it and instill 1 drop into the conjunctival sac of each eye, dropping them from above.
  Other Names: Control intervention
  Arms: Sodium Hyaluronate 0.18% (Vismed®)

SUMMARY:
This study aims at demonstrating the non-inferiority of Idroflog compared to sodium hyaluronate 0.18% for the disease improvement of people with documented history of dry eyes and use of tear substitutes for at least 3 months.

DETAILED DESCRIPTION:
This is a randomized, controlled, multicenter, assessor-blinded, non-inferiority trial comparing Idroflog® (sodium hyaluronate and hydrocortisone) with sodium hyaluronate in participants with dry eye disease (DED).

DED is a common, multifactorial ocular condition, which affects between 5% and 35% of adults worldwide and significantly affects their quality of life. DED treatment is based on the management of contributing factors (local environment, elimination of harmful systemic and topical drugs), eyelid hygiene and the use of artificial tears. The gold standard of the latter is sodium hyaluronate solutions, which, however, lack any anit-inflammatory activity necessary for DED's management. In comparison to these, Idroflog containing both sodium hyaluronate and hydrocortisone in addition to the usual activities of sodium hyaluronate artificial tears (diluent, diffusive, protective, nutrient, lubricant) also provides steroidal anti-inflammatory activity. Therefore, this study aims at showing that Idroflog® performs as well as current standard of care (sodium hyaluronate artificial tears) in the treatment of moderate DED, while providing a potential benefit on the control of the sub-clinical inflammatory component of DED and maintaining the excellent safety profile of sodium hyaluronate artificial tears treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged ≥ 18 years
* Documented history of dry eyes and use of tear substitutes for at least 3 months within the last year
* Presence of corneal fluorescein staining (Oxford Scale, Score ≥ 2) in at least one eye
* Ocular Surface Disease Index (OSDI) ≥ 23
* Reduced tear break-up time (< 11 seconds)

Exclusion Criteria:

* Women who are pregnant or lactating
* Best far corrected visual acuity < 1/10 in both eyes
* Known hypersensitivity to one of the components of the study medications or test products
* Use of any ocular topical medication other than the study medications for the treatment of ocular diseases including artificial tears during the study period
* Ocular surgery (of any type, including laser surgery and punctal plugs) or ocular trauma within the 4 months prior to screening
* Active ocular infection
* Active allergies requiring treatment
* Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in fluorescein corneal Staining (Oxford Scale 0-5) between inclusion and 30 days | 0 to 30 days of treatment

SECONDARY OUTCOMES:
Change From Baseline in fluorescein corneal Staining (Oxford Scale 0-5) between inclusion and 60 days, and between inclusion and 90 days. | 0 to 60 and 90 days of treatment
Change in OSDI between inclusion and 30, 60 and 90 days. | 0 to 30, 60 and 90 days of treatment
Change in Tear Film Break Up Time between inclusion and 30, 60 and 90 days | 0 to 30, 60 and 90 days of treatment
Change in Pentascore score between inclusion and 30, 60 and 90 days | 0 to 30, 60 and 90 days of treatment
Changes in Ocular Redness Scale (0-4; 0 = no ocular redness, 4 = extremely severe ocular redness) between inclusion and 30, 60 and 90 days | 0 to 30, 60 and 90 days of treatment
Safety 1: Changes in intraocular pressure between inclusion and 30, 60 and 90 days | 0 to 30, 60 and 90 days of treatment
Safety 2: Changes in visual acuity between inclusion and 90 days | 0 to 90 days of treatment

OTHER OUTCOMES:
Changes in non-specific inflammation markers (HLA-DR) at 30, 60 and 90 days in a subgroup of participants | 0 to 30, 60 and 90 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marc LABETOULLE, Pr., Principal Investigator — CHU Bicêtre, Service Ophtalmologie
Locations (5):
- France (5):
  - CHU Amiens-Picardie, Amiens
  - CHO Bordeaux - Site Pellegrin Centre François-Xavier Michelet, Service Ophtalmologie, Bordeaux
  - CHU Bicêtre, Service Ophtalmologie, Le Kremlin-Bicêtre
  - CHNO des 15-20, Paris
  - Hopital Fondation Adolphe de Rotschild, Paris

IPD SHARING:
Plan to Share IPD: Undecided
Results information from this trial will be submitted here to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 10 years after the completion of the primary endpoint by contacting the principal investigator, and upon authorization by the Sponsor.